CLINICAL TRIAL: NCT06302010
Title: The Effect of Stress Ball Intervention During Non-Stress Test on Anxiety and Fetal Well-Being in Women With High-risk Pregnancy: A Randomized Controlled Study
Brief Title: The Effect of Stress Ball Intervention During Non-Stress Test on Anxiety and Fetal Well-Being in High-Risk Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hümeyra TÜLEK DENİZ (Other)
Responsible Party: Sponsor-Investigator, Hümeyra TÜLEK DENİZ, Lecturer, Kafkas University
Organization: Kafkas University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KafkasU3636
Record Dates: First submitted 2024-02-10; First posted 2024-03-08 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-10

CONDITIONS: Anxiety; Fetal Conditions; Pregnancy Related
Keywords: anxiety; fetal well-being; high-risk pregnant women; Non stres test; stress ball; nurse
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The research will be conducted as a two-group, parallel, randomized, controlled experimental study with a pretest-posttest design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Pregnant women in the control group will not receive any intervention other than routine hospital care during the NST procedure.
- Intervention Group (Experimental): Pregnant women in the intervention group will be explained how to use the stress ball before NST. Pregnant women will be asked to demonstrate using a stress ball, and it will be verified that they can use it correctly. Pregnant women will be told to squeeze the ball once and release it after counting to three, to inhale each time they press the ball, to exhale when they relax their grip, and to focus only on the ball. Pregnant women will be instructed to continue this practice throughout the NST procedure (approximately 20 minutes). In addition, stress balls used in the hospital environment to minimize contamination will be disinfected with disposable asepsis wipes before being given to pregnant women.
  Interventions: Behavioral: Stress Ball Intervention

INTERVENTIONS:
Behavioral: Stress Ball Intervention — The stress ball has a soft plastic or silicone structure that can be held comfortably. Each ball is approximately 6 cm in diameter, in different colors, and is a soft toy that can be squeezed and manipulated with fingers to relieve stress and muscle tension and exercise the muscles (Apaydin Cirik et al., 2023). Squeezing a stress ball is a distraction and relaxation method. It is thought that squeezing a stress ball may be advantageous for reducing anxiety, considering its reliability, easy accessibility, effectiveness, low cost, sustainability, non-pharmacological and non-invasive properties.
  Arms: Intervention Group

SUMMARY:
This research will be conducted to determine the effect of stress ball intervention during NST on anxiety and fetal well-being in high-risk pregnant women. Women with high-risk pregnancies randomly assigned to intervention (n=43) and control (n=43) groups at a state and a faculty hospital in Turkey will be included in the study. Pregnant women in the intervention group will be told to squeeze and release the ball once after counting to three, to inhale each time they press the ball, to exhale when they relax their grip and to focus only on the ball. Pregnant women will be instructed to continue this practice throughout the NST procedure (approximately 20 minutes). Pregnant women in the control group will not receive any intervention other than routine hospital care during the NST procedure. Data on anxiety and fetal well-being outcomes will be collected before and after NST.

DETAILED DESCRIPTION:
Risky pregnancy refers to a situation in which there is a higher probability of negatively affecting the health and life of the pregnant woman and the fetus due to problems such as premature birth, premature rupture of membranes, cervical insufficiency, and placenta previa compared to normal pregnancies. Demographic and Health Research considers risky pregnancies as teenage pregnancies under the age of 18, pregnancies over the age of 35, births less than two years apart, and pregnancies with a parity of more than three births. Worldwide, 20 million women have high-risk pregnancies, and more than 800 women die from perinatal causes every day. 6-33% of these losses are in the high-risk pregnancy group. Worldwide, 5-10% of all pregnancies are complicated by preeclampsia. Malaria, tuberculosis, and chronic iron deficiency anemia are among the other most common pregnancy complications. In our country, the number of risky pregnancies has gradually decreased, but one in every three pregnant women is still a problematic pregnancy. Turkey Demographic and Health Surveys (TDHS) findings show that the risky pregnancy rate decreased from 44.3% to 35.2% in 25 years. According to the results of the 2014 Turkey Demographic and Health Surveys, the risky pregnancy rate, which was 31.1%, increased again in 2018.

In women who are diagnosed with complex and high-risk pregnancies that pose additional risks during pregnancy and have obstetric complications, the incidence of serious psychological problems, especially depression, is higher during pregnancy. The risk of anomaly diagnosed in the newborn causes maternal psychological issues throughout pregnancy. It has been shown that maternal psychosocial stress experienced during the antenatal period increases maternal infections, causes hormonal changes, and plays a role in the etiopathogenesis of fetal neurodevelopmental disorders, with long-term consequences such as poor birth outcomes including preterm birth and low birth weight, insulin resistance, and cardiovascular disease. High-risk pregnancies may require lifestyle changes, medical support, and even hospitalization. Depending on the severity of the pregnant woman's health condition, hospitalization may be necessary for high-risk pregnancies, starting weeks or months before the birth of the baby, and frequent NST monitoring may be required during this monitoring period. Risky pregnant women who are hospitalized during the antepartum period may experience psychological problems such as shock, depression, anxiety, sleep disorders, boredom, fear for the fetus and their health, guilt, feeling trapped, loss of control, weakness, loneliness, anger, and anxiety. The negative emotional state of a high-risk pregnant woman negatively affects the continuation of the pregnancy and may cause maternal-fetal attachment to be involved.

When biopsychosocial changes occur during pregnancy, maternal and fetal well-being must be maintained at the highest level. Nowadays, the Nonstress Test (NST) is widely used to evaluate fetal well-being in the intrauterine period because it is invasive and easy to interpret. NST is a non-invasive method with minimal risk for the mother and fetus, which is used to evaluate the fetal health status and maternal contractions in the prenatal period starting from the 32nd week of gestation and records the fetal heart rate with an electronic monitor. NST is based on the evaluation of fetal oxygenation. Although it is a painless procedure, it takes approximately 20 minutes, and the pregnant woman remains in the same position throughout the procedure, which creates stress and anxiety in the pregnant woman. High anxiety of the pregnant woman during the procedure affects the test result and may cause incorrect evaluation by increasing the false positivity rate. This increase in the false positivity rate in NST results may increase the practice of operative delivery.

It is the responsibility of nurses to eliminate situations that cause anxiety in pregnant women before and during the NST procedure and may affect the NST result. Stress ball, one of the non-pharmacological cognitive distraction methods, is easily accessible, low-cost, and reliable. When looking at the literature, the effects of the stress ball on psychometric parameters and vital signs such as anxiety, stress, depression, anxiety, comfort, and satisfaction in procedures such as colonoscopy, endoscopy, ESWL, prostate biopsy, radiography, hemodialysis, IV catheterization, PCR taking were examined. However, the effect of a stress ball on anxiety or the fetus during NST in high-risk pregnancies has not been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* Being over 18 years of age,
* Having a medically diagnosed risky condition during pregnancy (diabetes, hypertension, the threat of premature birth, eclampsia, etc.)
* Compliance with at least one of the criteria in the "Ministry of Health Pregnancy Risk Assessment Form" in the evaluation of "Current Pregnancy" (Table 1)
* Being at or above the 32nd week of pregnancy,
* Having a single living fetus,
* Having eaten at least two hours before the NST procedure,
* Not having smoked or consumed alcohol at least two hours before the NST procedure,
* Knowing how to read and write Turkish.

Exclusion Criteria:

* Deceleration or uterine contraction during NST,
* Presence of cardiovascular disease in the fetus,
* Presence of fetal distress,
* Presence of fetal anomaly,
* According to the physician, urgent intervention is needed,
* Having a diagnosed psychiatric disease,
* Having a visual, hearing, speaking, physical or mental disability.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 5 minutes before intervention and 5 minutes after the end of the intervention.
  The scale has 20 direct and reversed items, and each item is a 4-point Likert type. The total score from the scale varies between 20 and 80, with a higher score indicating a higher level of anxiety. Cronbach's alpha coefficient was 0.83 for State Anxiety.

SECONDARY OUTCOMES:
Fetal well-being | 5 minutes before the intervention and 5 minutes after the end of the intervention.
  This form was created based on the literature. As the secondary outcome measure of the research, fetal well-being will be recorded in this form.

CONTACTS AND LOCATIONS:
Overall Officials: Nazlı BALTACI, RN, PhD, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yilmaz D, Kutlu M, Baki E. A comparison of the effect on pain management of two non-pharmacological methods used during administration of Pfizer-BioNTech COVID-19 vaccine (BNT162b2): A randomized controlled study. Jpn J Nurs Sci. 2023 Jul;20(3):e12533. doi: 10.1111/jjns.12533. Epub 2023 Mar 31. PMID 36999594
- [Result] Yilmaz D, Gunes UY. The effect on pain of three different nonpharmacological methods in peripheral intravenous catheterisation in adults. J Clin Nurs. 2018 Mar;27(5-6):1073-1080. doi: 10.1111/jocn.14133. Epub 2018 Jan 8. PMID 29076581
- [Result] Hu HQ, Zhang J, Zhao W, Tian T, Huang AQ, Wang LL. [The occurrence and determinants of anxiety and depression symptoms in women of six counties/ districts in China during pregnancy]. Zhonghua Yu Fang Yi Xue Za Zhi. 2017 Jan 6;51(1):47-52. doi: 10.3760/cma.j.issn.0253-9624.2017.01.010. Chinese. PMID 28056270
- [Result] Quan X, Joseph A, Nanda U, Moyano-Smith O, Kanakri S, Ancheta C, Loveless EA. Improving Pediatric Radiography Patient Stress, Mood, and Parental Satisfaction Through Positive Environmental Distractions: A Randomized Control Trial. J Pediatr Nurs. 2016 Jan-Feb;31(1):e11-22. doi: 10.1016/j.pedn.2015.08.004. Epub 2015 Sep 26. PMID 26395650
- [Result] Ozen N, Berse S, Tosun B. Effects of using a stress ball on anxiety and depression in patients undergoing hemodialysis: A prospective, balanced, single-blind, crossover study. Hemodial Int. 2023 Oct;27(4):411-418. doi: 10.1111/hdi.13102. Epub 2023 Jun 15. PMID 37318078
- [Result] Gezginci E, Iyigun E, Yalcin S, Bedir S, Ozgok IY. Comparison of Two Different Distraction Methods Affecting the Level of Pain and Anxiety during Extracorporeal Shock Wave Lithotripsy: A Randomized Controlled Trial. Pain Manag Nurs. 2018 Jun;19(3):295-302. doi: 10.1016/j.pmn.2017.09.005. Epub 2017 Dec 14. PMID 29248604
- [Result] Gezginci E, Iyigun E, Kibar Y, Bedir S. Three Distraction Methods for Pain Reduction During Cystoscopy: A Randomized Controlled Trial Evaluating the Effects on Pain, Anxiety, and Satisfaction. J Endourol. 2018 Nov;32(11):1078-1084. doi: 10.1089/end.2018.0491. PMID 30280915
- [Result] Apaydin Cirik V, Turkmen AS, Ayaz M. Effectiveness of stress ball and relaxation exercises on polymerase chain reaction (RRT-PCR) test-induced fear and pain in adolescents in Turkiye. J Pediatr Nurs. 2023 Jul-Aug;71:135-140. doi: 10.1016/j.pedn.2022.12.001. Epub 2022 Dec 14. PMID 36526480
- [Result] Karatas TC, Gezginci E. The Effect of Using a Stress Ball During Endoscopy on Pain, Anxiety, and Satisfaction: A Randomized Controlled Trial. Gastroenterol Nurs. 2023 Jul-Aug 01;46(4):309-317. doi: 10.1097/SGA.0000000000000739. Epub 2023 May 17. PMID 37199436
- [Result] Kaasen A, Helbig A, Malt UF, Naes T, Skari H, Haugen G. Maternal psychological responses during pregnancy after ultrasonographic detection of structural fetal anomalies: A prospective longitudinal observational study. PLoS One. 2017 Mar 28;12(3):e0174412. doi: 10.1371/journal.pone.0174412. eCollection 2017. PMID 28350879
- [Result] Bolnick JM, Garcia G, Fletcher BG, Rayburn WF. Cross-over trial of fetal heart rate response to halogen light and vibroacoustic stimulation. J Matern Fetal Neonatal Med. 2006 Apr;19(4):215-9. doi: 10.1080/14767050500526131. PMID 16854694
- See also: HÜNEE (Hacettepe Üniversitesi Nüfus Etütler Enstitüsü). (2019). 2018 Türkiye nüfus ve Sağlık Araştırması. Hacettepe Üniversitesi Nüfus Etütler Enstitüsü, T.C. Cumhurbaşkanlığı Strateji ve Bütçe Başkanlığı ve TÜBİTAK, Ankara, Türkiye. — https://hips.hacettepe.edu.tr/tr/2018_turkiye_nufus_ve_saglik_arastirmasi-55
- See also: HÜNEE (Hacettepe Üniversitesi Nüfus Etütler Enstitüsü). (2014). 2014 Türkiye nüfus ve Sağlık Araştırması. Hacettepe Üniversitesi Nüfus Etütler Enstitüsü, T.C. Cumhurbaşkanlığı Strateji ve Bütçe Başkanlığı ve TÜBİTAK, Ankara, Türkiye. — https://hips.hacettepe.edu.tr/tr/2013_turkiye_nufus_ve_saglik_arastirmasi-67
- See also: HÜNEE (Hacettepe Üniversitesi Nüfus Etütler Enstitüsü). (1994). 1994 Türkiye nüfus ve Sağlık Araştırması. Hacettepe Üniversitesi Nüfus Etütler Enstitüsü, T.C. Cumhurbaşkanlığı Strateji ve Bütçe Başkanlığı ve TÜBİTAK, Ankara, Türkiye. — https://hips.hacettepe.edu.tr/tr/1993_turkiye_nufus_ve_saglik_arastirmasi-83
- See also: World Health Organization (WHO) (2018). Available from: Maternal mortality. Erişim Tarihi: 17.04.2023. — http://www.who.int/en/news-room/fact-sheets/detail/maternal-mortality